CLINICAL TRIAL: NCT02345434
Title: The Effect of Informative Letters on the Prescription and Receipt of Schedule II Controlled Substances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); General Services Administration (GSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JPAL-LETTERS-SII
Record Dates: First submitted 2014-10-06; First posted 2015-01-26 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Economics; Fraud; Delivery of Health Care; Health Expenditures; Centers for Medicare and Medicaid Services (U.S.)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No informative letter (No Intervention): This is the control arm and it involves no contact with the prescriber
- Informative letter (Experimental): This is the treatment arm; prescribers in this arm receive an informative letter (called a comparative billing report or peer activity report)
  Interventions: Other: Informative letter

INTERVENTIONS:
Other: Informative letter — The intervention is a letter that describes the Schedule II prescribing activity of the individual in comparison to a peer group of similar prescribers. It highlights the fact that the prescriber's activity is highly unlike her peers.
  Other Names: Comparative billing report; Peer activity report
  Arms: Informative letter

SUMMARY:
Fraud and waste is estimated to cost the American health care system nearly $200 billion each year, and the public Medicare and Medicaid programs about $60 billion each year. This study will evaluate a new method for fighting fraud: mailing informative letters to outlier providers to notify them of their aberrant behavior. These letters are targeted at high prescribers of schedule II controlled substances in Medicare Part D. The investigators will look at the effects of these letters on the behavior of providers and their patients. These effects are of substantial policy interest as they suggest how to best design anti-fraud policies. They are also of academic interest, shedding light on the behavior of physicians and their patients.

ELIGIBILITY:
Inclusion Criteria:

* Outlier with respect to the count of schedule II prescription drug events relative to peer group of prescribers in two of the three years 2011, 2012, and 2013
* Outlier with respect to the 30-day equivalent prescriptions of schedule II substances relative to peer group of prescribers in two of the three years 2011, 2012, and 2013

Exclusion Criteria:

- Deceased

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1525 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Finkelstein, PhD, Principal Investigator — Massachusetts Institute of Technology

REFERENCES:
- See also: American Economic Association Randomized Controlled Trials Registry Entry — https://www.socialscienceregistry.org/trials/525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no recruitment in the traditional sense. High prescribers of Schedule II controlled substances were identified in Medicare administrative data using a Tukey outlier method.
Pre-assignment Details: Seven of the identified outliers had died by the time of the study and were excluded from the intervention and later analysis.
Period: Overall Study
Arm/Group | No Informative Letter | Informative Letter
Started | 763 | 762
Completed | 758 | 760
Not Completed | 5 | 2
Not completed — Deceased (excluded from intervention and analysis) | 5 | 2

BASELINE CHARACTERISTICS:
Population: This baseline measure data was not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | No Informative Letter | Informative Letter | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years] — Population: Data for Baseline Measures were not collected
Sex: Female, Male — Population: Data for Baseline Measures were not collected
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 30-day Equivalent Prescribing of Schedule II Controlled Substances
Description: The prescribing of schedule II controlled substances over the 3 months following the initial sending of the letters. Prescribing is defined as the total "days supply" of schedule II controlled substances attributed to the prescriber, expressed in "30-day equivalents" i.e. divided by 30.
Time Frame: 3 months
Measure: Least Squares Mean (Standard Deviation); unit: 30-day equivalent prescription fills
Arm/Group | No Informative Letter | Informative Letter
Number analyzed (Participants) | 758 | 760
30-day equivalent prescription fills | 461.1 (443.9) | 450.0 (450.9)
Statistical Analysis 1: Comparison: No Informative Letter vs Informative Letter; Test type: Superiority; Mean Difference (Final Values) = 3.53, 95% CI 2-sided [-6.35 to 13.4]

2. Secondary Outcome: 30-day Equivalent Prescribing of Schedule II Controlled Substances
Time Frame: 1 month
Measure: Least Squares Mean (Standard Deviation); unit: 30-day equivalent prescription fills
Arm/Group | No Informative Letter | Informative Letter
Number analyzed (Participants) | 758 | 760
30-day equivalent prescription fills | 155.5 (148.8) | 151.1 (150.4)
Statistical Analysis 1: Comparison: No Informative Letter vs Informative Letter; Test type: Superiority; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-3.68 to 2.1]

3. Secondary Outcome: 30-day Equivalent Prescribing of Schedule II Controlled Substances
Time Frame: 6 months
Population: Outcome measure not collected for study
Arm/Group | No Informative Letter | Informative Letter
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: 30-day Equivalent Prescribing of Schedule II Controlled Substances
Time Frame: 9 months
Population: Outcome measure not collected for study
Arm/Group | No Informative Letter | Informative Letter
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 30-day Equivalent Prescribing of Schedule II Controlled Substances
Time Frame: 1 year
Population: Outcome measure not collected for study
Arm/Group | No Informative Letter | Informative Letter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | No Informative Letter | Informative Letter
Serious Adverse Events (participants affected / at risk) | 0/758 | 0/760
Other Adverse Events (participants affected / at risk) | 0/758 | 0/760

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No